CLINICAL TRIAL: NCT05975853
Title: Examining the Effects of Binaural Beat Music on Sleep Quality, Heart Rate Variability, and Depression in Older People With Poor Sleep Quality in a Long-term Care Institution: A Randomized Controlled Trial
Brief Title: Effects of Binaural Beat Music on Elderly Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Yang Shang-Yu, Assistant professor, Asia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Asia0727
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Sleep Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Binaural beat music group (BBM group) (Experimental): 20 minutes of music thrice a week (Monday, Wednesday, and Friday) for two weeks (total of 12 times)
  Interventions: Other: Binaural beat music group (BBM group)
- Control group (Sham Comparator): 20 minutes of music thrice a week (Monday, Wednesday, and Friday) for two weeks (total of 12 times)
  Interventions: Other: Control group

INTERVENTIONS:
Other: Binaural beat music group (BBM group) — The participant sat on a chair with eyes closed and wore over-ear stereo headphones to listen to 15 minutes of Taiwanese Hokkien oldies (familiar music, can be selected by participant) with BBM embedded.
  Arms: Binaural beat music group (BBM group)
Other: Control group — The participant sat on a chair with eyes closed and wore over-ear stereo headphones to listen to 15 minutes of Taiwanese Hokkien oldies (familiar music, can be selected by participant) without BBM embedded.
  Arms: Control group

SUMMARY:
Background:

Older people in long-term care institutions often have poor sleep quality and depression, which may negatively affect their health and welfare. Binaural beat music (BBM) has been proposed as a possible intervention. However, its effects on older people with poor sleep quality in long-term care institutions is still unclear.

Objective:

This study aimed to examine the effects of binaural beat music on sleep quality, heart rate variability, and depression in older people with poor sleep quality in a long-term care institution

Methods:

A single-blind randomized controlled trial design was employed and 64 older participants with poor sleep quality were recruited from a long-term care institution in Taiwan. Participants were randomized into the BBM group or control (sham) group (32 per group) and received 14 days of intervention. During the intervention period, participants in the experimental group listened to 20 minutes of Taiwanese Hokkien oldies embedded with BBM once in the morning and afternoon thrice a week. Participants in the control group only listened to Taiwanese Hokkien oldies. Questionnaires and heart rate variability analysis were used to assess participants' sleep quality, heart rate variability, and depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were participants who: were aged 65 years and older, had a PSQI score> 7, were able to understand questionnaire contents and communicate in Mandarin or Taiwanese Hokkien, stayed in institution for 1 month and more, and did not receive antidepressant within 3 months prior to and during the intervention.

Exclusion Criteria:

* Exclusion criteria were those with hearing loss, history of bipolar disorder or schizophrenia diagnosed by a physician, and had an acute physiological disease, such as cold, fracture, or trauma.

Ages: 75 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | On Day 14 of the intervention, the researchers conducted the posttest (second test) at the participants' long-term care institution and the test content was the same as the first test. It took about 10 minutes.
  There were 18 questions in the PSQI, and participants used a self-rated method to fill in their sleep quality in the last month on a 4-point Likert scale. The total score range was 0-21 points. The higher the score, the poorer the sleep quality. This scale has seven dimensions, including: (1) Subjective sleep quality; (2) Sleep latency; (3) Sleep duration; (4) Sleep efficiency; (5) Sleep disturbances; (6) Daytime dysfunction; and (7) Use of sleep medication. PSQI had good validity and reliability(Tsai et al., 2005).
HRV analyzer | On Day 14 of the intervention, the researchers conducted the posttest (second test) at the participants' long-term care institution and the test content was the same as the first test. It took about 5 minutes
  HRV was used to measure heart rate variability, including five markers: (1) Mean heart rate; (2) SDNN: Standard deviation of all RR intervals, represent the physiological health of autonomic nervous system; the higher the SDNN, the better the physiological health of the autonomic nervous system; (3) nLF: Normalized low frequency, reflects sympathetic nervous activity. The higher the value, the greater the activity; (4) nHF: Normalized high frequency, reflects parasympathetic nervous activity. The higher the value, the greater the activity; (5) LF/HF, a marker reflecting sympathetic and parasympathetic nervous activity.

SECONDARY OUTCOMES:
Geriatric Depression Scale (GDS) | On Day 14 of the intervention, the researchers conducted the posttest (second test) at the participants' long-term care institution and the test content was the same as the first test. It took about 5 minutes
  The GDS was a self-rated scale used to evaluate depression status in older people. This scale contained 30 questions and a binary scoring method (Yes/No). We used the 15-item version and the total score ranged from 0 to 15 points. Scores of 0-4, 5-8, 9-11, and 12-15 points indicated normal, mild, moderate, and severe depression, respectively. A higher total score indicated greater depression severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Asia Univeraity, Taichung, WuFeng, Taiwan